CLINICAL TRIAL: NCT05737030
Title: An Observational Study on the Effect of L-ornithine-L-aspertate (LOLA) on the Flavonifractor Abundance in the Gut Microbiome in Liver Cirrhosis
Brief Title: Effect of L-ornithine-L-aspertate (LOLA) on the Gut Microbiome
Acronym: LOLAbiome
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: CBmed Ges.m.b.H. (Other)
Responsible Party: Principal Investigator, Vanessa Stadlbauer-Koellner, MD, Principal investigator, Medical University of Graz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOLAbiome; 2022-002924-11 (EudraCT Number)
Record Dates: First submitted 2023-02-12; First posted 2023-02-21 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — ornithylaspartate; Silybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- L-ornithine-L-aspertate (Experimental): L-ornithine-L-aspertate 18g per day
  Interventions: Drug: L-ornithine L-aspartate

INTERVENTIONS:
Drug: L-ornithine L-aspartate — Amino acid combination
  Other Names: Hepa-Merz

SUMMARY:
Study to test the effect of the drug "L-ornithine.L-aspertate" (LOLA) on microorganisms in the digestive tract in patients with liver cirrhosis (damage of the liver due to liver disease)

DETAILED DESCRIPTION:
Liver cirrhosis is associated with gut microbiome dysbiosis, which may drive intestinal inflammation, gut barrier dysfunction and the development of complications. LOLA is a well-established drug against elevated ammonia levels that contribute to hepatic encephalopathy and sarcopenia. In a recent retrospective study, LOLA has been shown to improve gut microbiome dysbiosis.

In this study we aim to investigate whether LOLA therapy over three months in patients with liver cirrhosis (irrespective of the etiology) and covert or overt hepatic encephalopathy (HE) leads to an improvement in gut microbiome dysbiosis, as well as markers of gut permeability, inflammation, muscle function and ammonia levels.

ELIGIBILITY:
Inclusion Criteria:

* • Liver cirrhosis (clinical/radiological/histological diagnosis)

  * Indication for LOLA use (covert or over hepatic encephalopathy, Grad 0-2))
  * Written informed consent
  * Age 18 -100 years

Exclusion Criteria:

* • Allergy to LOLA or its constituents, or to medications with a similar chemical structure (oral nutritional supplements are allowed when stable >/= 8 weeks before and during the study)

  * Recent (</= 8 weeks) changes of the dose of the lactulose therapy for hepatic encephalopathy
  * Rifaximin or any other antibiotic therapy within the past 4 weeks
  * Intake of LOLA in the past four weeks before inclusion
  * Intake of L-dopamine
  * Renal insufficiency with a serum creatinine >3mg/dl
  * Hepatocellular carcinoma BCLC D under best supportive care
  * Inability to give informed consent
  * Pregnancy or breastfeeding
  * Participation in another interventional trial within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Microbiome | 3 months
  Increase of the genus Flavonifractor in the gut microbiome after 3 months of LOLA treatment

SECONDARY OUTCOMES:
Alpha diversity | 3 months
  Change in alpha diversity of the gut microbiome after 3 months of LOLA treatment
Beta diversity | 3 months
  Change in beta diversity of the gut microbiome after 3 months of LOLA treatment
Taxonomic composition | 3 months
  Change in taxonomic composition (beyond Flavonifractor) of the gut microbiome after 3 months of LOLA treatment
Predicted metagenomics | 3 months
  Change in predicted gut microbiome function after 3 months of LOLA treatment
Metabolomics | 3 months
  Change in stool, serum or urine metabolite composition after 3 months of LOLA treatment
Gut permeability | 3 months
  Change in biomarkers of gut permeability (zonulin, DAO, sCD14, LBP) after 3 months of LOLA treatment
Handgrip strength | 3 months
  Change in handgrip strength after 3 months of LOLA treatment
Muscle function | 3 months
  Change in gait speed and balance after 3 months of LOLA treatment
Ammonia in serum | 3 months
  Change in ammonia blood levels after 3 months of LOLA treatment
Mid-arm circumference and triceps fold thickness | 3 months
  Change in anthropometric parameters (Mid-arm circumference and triceps fold thickness) after 3 months of LOLA treatment
short form (SF)-36 | 3 months
  Change in quality of life after 3 months of LOLA treatment, 8 domains, 0-100 points, higher points indicate higher quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
Sequencing data will be deposited in an open access repository together with metadata
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2023
Access Criteria: open access

REFERENCES:
- [Derived] Habich D, Horvath A, Feldbacher N, Rebol L, Nepel M, Madl T, Habisch HJ, Baumann-Durchschein F, Furst S, Plank J, Rainer F, Spindelbock W, Stauber RE, Tatscher E, Wagner M, Zollner G, Stadlbauer V. An observational study on the effect of l-ornithine-l-aspartate (LOLA) on the gut microbiome in liver cirrhosis. A single center phase 4 study. Clin Nutr. 2025 Nov 29;56:106522. doi: 10.1016/j.clnu.2025.11.007. Online ahead of print. PMID 41406626